CLINICAL TRIAL: NCT06462664
Title: Exploring the Impact of Monocytes in Myeloproliferative Neoplasia
Brief Title: Exploring the Impact of Monocytes in Myeloproliferative Neoplasia (EMYNEM)
Acronym: EMYNEM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0134 - EMYNEM
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Impact of monocytes on Myeloproliferative Neoplasm hematopoietic stem cell growth and differentiation in vitro

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MPN in the participating center
* Over 18 yo

Exclusion Criteria:

* Not able to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with MPN
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Proliferation and differentiation of hematopoitic stem/progenitor cells | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement